CLINICAL TRIAL: NCT00128778
Title: Phase IV.III Clinical Trial to Evaluate Maintenance Treatment With Caelyx vs. Observation After Administration of Induction Chemotherapy in Metastatic Breast Cancer Patients
Brief Title: Maintenance Treatment With Liposomal Doxorubicin (Caelyx) in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 2001-01
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; Metastases; Maintenance treatment
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — liposomal doxorubicin

ARMS (2):
- Arm A: PLD (Experimental): Pegylated liposomal doxorubicin (PLD) after induction chemotherapy in patients with metastatic breast cancer (MBC). Patients without disease progression following first-line induction chemotherapy consisting of three cycles of doxorubicin (75 mg/m2) followed by three cycles of docetaxel (100 mg/m2) both every 21 days, were randomized to PLD (40 mg/m2) every 28 days for six cycles or to observation.
  Interventions: Drug: Pegylated liposomal doxorubicin
- Arm B: Observation (No Intervention): Patients without disease progression following first-line induction chemotherapy consisting of three cycles of doxorubicin (75 mg/m2) followed by three cycles of docetaxel (100 mg/m2) both every 21 days, were randomized to observation.

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin
  Other Names: Caelyx
  Arms: Arm A: PLD

SUMMARY:
This is a randomized, prospective and multicenter phase IV clinical trial, which has been designed as a phase III study. One hundred fifty-four women (77 per treatment arm) will be recruited in the study.

DETAILED DESCRIPTION:
The main variable is time to disease progression. All patients must be treated with first line of induction chemotherapy, consisting of doxorubicin 75 mg/m2, day 1 every 3 weeks, and docetaxel, 100 mg/m2, day 1 every 3 weeks. Both drugs must be administered sequentially. Patients previously treated with anthracyclines must receive 2 courses of doxorubicin and 4 courses of docetaxel. Otherwise, patients will receive 3 courses of doxorubicin followed by 3 courses of docetaxel.

Patients with complete response, partial response or stable disease are eligible for 2001-01 study.

The investigators assume that maintenance treatment with Caelyx will increase mean time to progression from 10, 46 months (observation) to 17, 43 months. Expected difference in mean time to progression is 6, 97 months (Hazard ratio = 0.6). With an alpha error of 0.01 (unilateral) and power of 80%, 77 patients per arm are needed, 154 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients with metastatic breast cancer who have responded to a first line induction chemotherapy treatment.
* Age: at least 18 years old.
* Performance status Eastern Cooperative Oncology Group (ECOG) scale 0, 1, 2.
* Normal cardiac function, confirmed by left ventricular ejection fraction (LVEF).
* Hematology: leucocytes >= 4 x 10^9/l; neutrophils >= 2.0 x 10^9/l; platelets >= 100 x 10^9/l; hemoglobin <= 10 g/dl.
* Hepatic function: total bilirubin < 1 upper limit of normal (UNL); aspartate aminotransferase (ASAT) (SGOT) and alanine aminotransferase (ALAT) (SGPT) < 2.5 UNL; alkaline phosphatase < 5 UNL. Patients with ASAT (SGOT) and ALAT (SGPT) > 1.5 UNL and alkaline phosphatase > 2.5 UNL are not eligible.
* Renal function: creatinine < 175 mmol/l (2 mg/dl); creatinine clearance > 45 ml/min.

Exclusion Criteria:

* Pregnant or lactating patients.
* Previous cardiac dysfunction grade II or higher as per New York Heart Association, along with congestive cardiac failure.
* Hypersensitivity to anthracyclines or Cremophor®.
* Clinically significant hepatic dysfunction.
* Current uncontrolled infection.
* Mental confusion and lack of orientation.
* Any circumstance precluding an adequate follow-up.
* Radiotherapy in the previous 4 weeks.
* Any other concurrent neoplasm, except for basal cell carcinoma or in situ carcinoma.
* Symptomatic metastasis in the brain.
* Previous radiotherapy radiating a third of haematopoietic centres.
* Males.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2002-10-28 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2010-07-07 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | Through study completion, an average of 1 year
  Tumor assessments will be performed until disease progression in order to evaluate the TTP. TTP is defined as the time from the date of the first dose to the first date of objectively determined progressive disease. For patients not known to have objectively-determined progressive disease, TTP will be censored at the date of the last objective progression-free assessment. For patients who receive subsequent systemic anticancer therapy (after discontinuation from the study treatment) prior to objective disease progression, TTP will be censored at the date of last objective progression-free assessment prior to the initiation of postdiscontinuation systemic anticancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Universitario Virgen de la Victoria
Locations (1):
- Spanish Breast Cancer Research Group (GEICAM), San Sebastián de los Reyes, Madrid, Spain

REFERENCES:
- [Result] Alba E, Ruiz-Borrego M, Margeli M, Rodriguez-Lescure A, Sanchez-Rovira P, Ruiz A, Mel-Lorenzo JR, Ramos-Vazquez M, Ribelles N, Calvo E, Casado A, Marquez A, Vicente D, Garcia-Saenz JA, Martin M. Maintenance treatment with pegylated liposomal doxorubicin versus observation following induction chemotherapy for metastatic breast cancer: GEICAM 2001-01 study. Breast Cancer Res Treat. 2010 Jul;122(1):169-76. doi: 10.1007/s10549-010-0860-9. Epub 2010 Apr 2. PMID 20361253
- See also: Click here for more information about this study — http://www.geicam.org